CLINICAL TRIAL: NCT02249221
Title: A Randomized (Part B), Open-label (Part A) or Double-blind (Part B), Active-controlled (Part B) Phase I/IIa Study to Investigate the Safety, Tolerability, and Immunogenicity of GC3106 (Quadrivalent Cell-culture Based Influenza Vaccine)
Brief Title: Safety, Tolerability, and Immunogenicity of GC3106 (Quadrivalent Cell-culture Based Influenza Vaccine)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GC3106_P1/2a
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Influenza
Keywords: Influenza vaccine; Vaccination; cell-culture based influenza vaccine; cell culture derived influenza vaccine; CCIV
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quadrivalent cell-culture based influenza vaccin (Experimental): Day 1: GC3106, 0.5ml, intramuscular, a single dosing
  Interventions: Biological: Quadrivalent cell-culture based influenza vaccin
- Trivalent influenza vaccine (Active Comparator): Day 1: GC Flu Pre-filled Syringe Inj., 0.5ml, intramuscular, a single dosing
  Interventions: Biological: Trivalent influenza vaccine

INTERVENTIONS:
Biological: Quadrivalent cell-culture based influenza vaccin — GC3106, 0.5ml, intramuscular, a single dosing at Day 1
  Other Names: GC3106
  Arms: Quadrivalent cell-culture based influenza vaccin
Biological: Trivalent influenza vaccine — GC Flu Pre-filled Syringe Inj., 0.5ml, intramuscular, a single dosing at Day 1
  Other Names: GC Flu Pre-filled Syringe Inj.
  Arms: Trivalent influenza vaccine

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and immunogenicity of GC3106 after single intramuscular administration in Korean healthy adults.

DETAILED DESCRIPTION:
This study is the first in human trial of GC3106 and is designed as an adaptive Phase I/IIa to ensure participants protection. Part A is an open-label and single arm study in 9 healthy volunteers. Data and Safety Monitoring Board (DSMB) will review the solicited/unsolicited adverse events conditionally if any toxicity of Grade 3 or 4 has been reported during 7 days after vaccination from the first 9 healthy volunteers. Part B is a randomized (2:1), double-blind, active controlled study and a total of 75 volunteers will participate in this part. Adverse events assessment will be done according to the 'Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials'.

ELIGIBILITY:
Inclusion Criteria:

* Given written informed consent
* Healthy Korean adults (age: between over 19 and under 65)
* Korean adults who agree with 21 days follow up after vaccination and good compliance to study procedures
* Those who are able to comply with the requirements for the study

Exclusion Criteria:

* Inability in written/verbal communication
* Subjects who have participated in other interventional study within 30 days
* Alcohol or drug abuse within 6 months
* Heavy drinkers or subjects who do not agree to stop drinking for 3 days before vaccination and other 3 days after vaccination
* Who got the treatment of psychotropic drugs and narcotic analgesic drugs within 6 months of enrollment
* Hypersensitivity with drug or active ingredient
* Disorders in immune function
* History of Guillain-Barré syndrome
* Disease/medications which are likely to cause any severe bleeding
* Active infection or experience of fever (>38.0 ℃) within 72 hours following vaccination
* Oral temperature >38.0 ℃ at the vaccination day
* Erythema, tattoo, injury at shoulder (vaccination site)
* Influenza vaccination within 6months
* Any vaccination within 30 days
* Concomitant medications/therapy such as immunosuppressants or immune modifying drugs, systemic corticosteroids, immunoglobulins, blood or blood- derived products, or anti-cancer chemotherapy or radiation therapy within3 months
* Pregnant or breast-feeding women
* Clinically significant underlying diseases or medical history at investigator's discretion

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Solicited adverse events following vaccination | Day 1 up to 7 Days post vaccination
  Solicited injection site reactions: Pain, Tenderness, Erythema, Redness, Induration, and Swelling; Solicited systemic reactions: Fever, Sweating, Chill, Nausea, Vomiting, Diarrhea, Headache, Fatigue, Myalgia, arthralgia.
Unsolicited adverse events following vaccination | Day 1 up to 22 Days post vaccination
  It can be estimated by Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials
Abnormalities in physical examination, vital signs, and/or clinical laboratory tests | Day 22 post vaccination

SECONDARY OUTCOMES:
Seroprotection rate of HI (Hemagglutination Inhibition) antibody for each strain | Day 22 post vaccination
Seroconversion rate of HI (Hemagglutination Inhibition) antibody for each strain | Day 22 post vaccination
GMT(geometric mean titers) for each strain | Day 22 post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Woo Joo KIM, M.D., Ph.D, Principal Investigator — Korea University Guro Hospital; Chang-Hee LEE, M.D., Study Director — Green Cross Corporation
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea